CLINICAL TRIAL: NCT01605591
Title: Comparison of Different Bending Mode for Double-lumen Endotracheal Tube Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUH-IRB-20110172
Record Dates: First submitted 2011-10-16; First posted 2012-05-25 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia Intubation Complications
Keywords: left-side double lumen bronchial tube; bending type; GlideScope videolaryngoscope

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the DLT bending to the right (Active Comparator)
  Interventions: Procedure: the DLT bending to the right
- the DLT bending to the left (Active Comparator)
  Interventions: Procedure: the DLT bending to the left

INTERVENTIONS:
Procedure: the DLT bending to the right — bending the bronchial lumen of DLT 60~90 degrees in the same side with the tracheal lumen
  Other Names: different bending mode of DLT
  Arms: the DLT bending to the right
Procedure: the DLT bending to the left — bending the bronchial lumen of DLT 60~90 degree opposed to the tracheal lumen
  Other Names: different bending mode of DLT
  Arms: the DLT bending to the left

SUMMARY:
The purpose of this study is to comparing the effects of different double-lumen endotracheal tube's bending type in tracheal intubation.

DETAILED DESCRIPTION:
Intubation with the double-lumen endotracheal tube (DLT) remains a great challenge for anesthesiologists. Although new upper airway devices, such as GlideScope(R) videolaryngoscope, had been developed for facilitating airway management, the larger size and the complexity of DLT than single-lumen tube (SLT) makes the difficulties for DLT intubation. Therefore, the investigators designed this study to investigate the effects of different bending type of DLT in tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status I-III
2. more than 18 years of age
3. Receiving thoracic surgery with double-lumen endobronchial tube

Exclusion Criteria:

1. risk of regurgitation and pulmonary aspiration
2. history of gastroesophageal reflux
3. pregnancy
4. scheduled tracheostomy and postoperative prolonged ventilation in ICU
5. limited neck extension (< 35°)
6. a thyromental distance less than 7 cm
7. a sternomental distance less than 12.5 cm with the head fully extended
8. mouth can not open

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Main outcome measure is the successful rate of the first intubation compared with the two bending modes of DLT | 12 month

SECONDARY OUTCOMES:
the time needed to insert the DLT during the period of intubation | 12 months
mean blood pressure (MAP) before intubation, and after intubation 1, 3,and 5 min | 12 months
the incidence of hypoxemia during the period of intubation | 12 months
  Hypoxemia is defined as the SPO2 is below 90%.
the heart rate (HR) before intubation, and after intubation 1, 3,and 5 min | 12 months
the incidence of sore throat after extubation | 12 months
the incidence of hoarseness after extubation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, VS, Principal Investigator — Department of anesthesia, Kaoshiung medical university hospital
Locations (1):
- department of anesthesia, Kaohsiung medical university memorial hospital, Kaohsiung City, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Hsu HT, Chou SH, Chou CY, Tseng KY, Kuo YW, Chen MC, Cheng KI. A modified technique to improve the outcome of intubation with a left-sided double-lumen endobronchial tube. BMC Anesthesiol. 2014 Aug 18;14:72. doi: 10.1186/1471-2253-14-72. eCollection 2014. PMID 25206313